CLINICAL TRIAL: NCT03417882
Title: A Pilot, Open-Label, Multi-Center, Multi-Dose Study of GRN-1201 Added to Pembrolizumab in Subjects With Non-Small Cell Lung Cancer With High PD-L1 Expression
Brief Title: GRN-1201 With Pembrolizumab in Subjects With Metastatic PD-L1+ NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment rate too slow
Sponsor: BrightPath Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRN-1201-002
Record Dates: First submitted 2017-11-14; First posted 2018-01-31 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Metastatic NSCLC
Keywords: PD-L1+
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The study will follow a Simon two-stage design [1] with up to 64 subjects enrolled. All subjects will receive GRN-1201 at a dose of 3.0 mg per peptide in combination with 75 µg sargramostim (Leukine®) and 200 mg pembrolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): All subjects will have newly diagnosed, metastatic PD-L1+ (TPS ≥ 50%) NSCLC with no epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations.
  Interventions: Biological: GRN-1201 + Pembrolizumab

INTERVENTIONS:
Biological: GRN-1201 + Pembrolizumab — GRN-1201 will be administered in combination with Pembrolizumab
  Other Names: Pembrolizumab

SUMMARY:
This is a non-randomized, Phase 2, 2-stage, open-label, multi-center study of GRN-1201/sargramostim + pembrolizumab in subjects with PD-L1+ metastatic NSCLC. All subjects will have newly diagnosed metastatic PD-L1+ (TPS ≥ 50%) NSCLC with no epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations. Subjects with EGFR or ALK genomic tumor aberrations with progression on FDA-approved therapy for these aberrations are eligible

DETAILED DESCRIPTION:
This is a non-randomized, Phase 2, 2-stage, open-label, multi-center study of GRN-1201/sargramostim + pembrolizumab in subjects with metastatic PD-L1+ NSCLC.

All subjects will have newly diagnosed metastatic PD-L1+ (TPS ≥ 50%) NSCLC with no epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations.

The study will follow a Simon two-stage design with up to 64 total subjects enrolled. All subjects will receive GRN-1201 at 3.0 mg in combination with 75 µg sargramostim and 200 mg pembrolizumab.

GRN-1201 is to be administered once weekly for 4 weeks followed by every 3-week dosing for an additional 12 doses (16 total doses of GRN-1201). Each dose of GRN-1201 will be given as 1 mL divided into 4 separate 0.25 mL intradermal injections on each day of treatment. Pembrolizumab is to be given every 3 weeks for up to a total of 35 doses.

This study will consist of a screening period of up to 28 days; a treatment period consisting of GRN-1201/sargramostim administered weekly for 4 weeks (4 doses) followed by administration every 3 weeks for 12 additional doses . Pembrolizumab is to be given every 3 weeks for up to a total of 35 doses.

A follow up visit will occur approximately 4 weeks after the last administration of treatment for the study. In addition, all subjects will be followed for evaluation of disease progression and survival

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female at least 18 years of age (at the time consent is obtained);
2. Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures);
3. Have histologically- or cytologically-confirmed diagnosis of Stage IV NSCLC Have newly diagnosed, metastatic NSCLC with PD-L1 TPS ≥ 50% (as determined by central lab using the 22C3 pharmDx kit) Note: Subjects with documentation of PD-L1 TPS ≥50% by IHC analysis using the 22C3 pharmDx kit will not require repeat PD-L1 testing by central laboratory and
4. Have no prior systemic chemotherapy for metastatic disease: at least 6 months since prior adjuvant chemotherapy
5. Be HLA-A*02+ as determined by Central Laboratory;
6. Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy;
7. Have a life expectancy of at least 3 months;
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
9. Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team. Target tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions;
10. Has adequate organ function as defined by:

    * Absolute neutrophil count ≥ 1,500/µL
    * Platelets ≥ 100,000/µL
    * Hemoglobin ≥ 9 g/dL (without transfusion for at least one month)
    * Serum creatinine ≤ 1.5 x Upper Limit of Normal (ULN) OR

      o glomerular filtration rate (GFR) ≥30mL/min if serum creatinine > 1.5 x ULN, creatinine clearance may be calculated using the institutional/laboratory standard method
    * Serum total bilirubin ≤ 1.5 x ULN OR

      o Direct bilirubin ≤ ULN for subjects with total bilirubin >1.5 x ULN
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver metastases)
    * Albumin ≥2.5mg/dL
    * International Normalized Ratio (INR) or PT/aPTT <1.5 x ULN. For subjects receiving anticoagulation therapy, PT/aPTT and INR should not be greater than the recommended range for the intended use of the anticoagulant
11. Have recovered from the effects of any prior radiotherapy or surgery;
12. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropic (hCG) test within 1 week of Day 1 (pregnancy test not required for subjects with bilateral oophorectomy and/or hysterectomy or for those subjects who are >1 year post-menopausal); and
13. All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 4 months after the last dose of study treatment.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 14 days of the first dose of treatment;
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 10 mg prednisone or equivalent per day or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment;
3. Has undergone major surgery within 3 weeks of Study Day 1, Subject must have recovered adequately from any toxicity and/or complications from the intervention prior to starting therapy;
4. Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], GM-CSF or recombinant erythropoietin) within 4 weeks prior to study Day 1;
6. Has known active central nervous system (CNS) metastases NOTE: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either magnetic resonance imaging (MRI) or computerized tomography (CT) scan] for at least four weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment;
7. Has carcinomatous meningitis;
8. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study;
9. Has history of interstitial lung disease, or history of (non-infectious) pneumonitis that required steroids, or current pneumonitis;
10. Has an active infection requiring systemic therapy NOTE: Antibiotic therapy must have been completed a minimum of 3 days prior to start of study treatment;
11. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
12. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to day 1 of study treatment;
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator;
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study;
15. Has received a live virus vaccine within 30 days of the planned first dose of study therapy NOTE: seasonal influenza vaccines for injection which are generally inactivated flu vaccines are permitted; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not permitted;
16. Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment; or
17. Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.
18. Have an EGFR or ALK genomic tumor aberrations for which targeted therapy with an EGFR or ALK inhibitor is indicated.

    Additional Exclusion Criteria for Cohort 2:
19. Has had prior treatment with an anti-PD-1 or anti-PD-L1 antibody, anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab) or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Assess the effect, as measured by response rate of the addition of GRN-1201 to Pembrolizumab | First dose through 16 weeks after last dose of study drug
  Tumor assessment over time using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

SECONDARY OUTCOMES:
Evaluate the adverse event profile for the combination of GRN-1201 and Pembrolizumab as assessed by treatment -related events according to CTCAE version 4 | First dose through 16 weeks after last dose of study drug
  The safety and tolerability of GRN-1201/sargramostim + pembrolizumab will be evaluated by local and systemic signs and symptoms of injection site reactions, and incidence of adverse events including immune related adverse events (irAEs).
Host immune response to GRN-1201 | First dose through 16 weeks after last dose of study drug
  Immune responses to GRN-1201 will be monitored to establish proof-of principle for the proposed pharmacological effect and demonstrate immunogenicity of GRN-1201.
  Immune response to the individual peptides will be assessed by measurement of cytotoxic T lymphocytes (CTLs) (by gamma interferon [IFN-γ] ELISPOT assay) and by measurement of antibodies to each peptide
Clinical Benefit response rate (CR + PR + SD >/= 16 weeks) | First dose through 16 weeks after last dose of study drug
  Tumor assessment over time using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Progression-free survival | First dose through 2 years after last dose of combination treatment
  Progression-free survival will be determined by tumor assessments or death from any cause
Duration of response in responding subjects | First dose through 16 weeks after last dose of study drug
  The duration of objective response will be assessed
Duration of clinical benefit | First dose through 16 weeks after last dose of study drug
  The duration of clinical benefit response rate will be assessed
Overall survival | First dose through 16 weeks after last dose of study drug
  All subjects will be followed for overall survival after discontinuation of combination treatment

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - St Joseph Hospital of Orange, Orange, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Florida Hosptial Cancer Center- AdventHealth, Orlando, Florida
  - Robert H Lurie Cancer Center at Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Orchard Healthcare, Skokie, Illinois
  - Norton Healthcare Cancer Institute, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Ocshner Cancer Institute, New Orleans, Louisiana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Virginia Cancer Institute, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided